CLINICAL TRIAL: NCT01091753
Title: Effect of Nocturnal Administration of Anti-hypertensive Medications in NoN-dippers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Choi, Dong hun/professor, Yonsei University, College of Medicine
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 4-2007-0440
Record Dates: First submitted 2010-03-23; First posted 2010-03-24 (Estimated); Last update posted 2010-10-08 (Estimated); Status verified 2010-10

CONDITIONS: Hypertension
Keywords: Non-dipper HTN patient
MeSH Terms: conditions — Hypertension | interventions — Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- morning administration group (Placebo Comparator)
  Interventions: Drug: Valsaltan, amlodipine
- nocturnal administration group (Experimental)
  Interventions: Drug: Valsaltan, amlodipine

INTERVENTIONS:
Drug: Valsaltan, amlodipine — nti hypertensive medication time (nocturnal administration vs morning administration

SUMMARY:
The purpose of this study is to determine the effect of nocturnal administration of Anti-hypertensive medications in Non-dippers.

Efficacy variables.

1. ECHO
2. 24hr. horter
3. IMT
4. BUN/crea, urine analysis (microalbulinuria
5. Cardio vascular event. "

ELIGIBILITY:
Inclusion Criteria:

1. Essential hypertension (stage 1-2)
2. 24hr. holer : non-dipper
3. Age 18 ~70.

Exclusion Criteria:

1. Any known malignant disease
2. Renal failure , creatinine >2.0mg/dl
3. Liver disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-03; Primary Completion 2009-05 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
IMT(intima media thickness) Measure data(Sono) | baseline
IMT(intima media thickness) Measure data(Sono) | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Dong hun Choi, Principal Investigator — professor of division of Cardiology
Locations (1):
- Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea